CLINICAL TRIAL: NCT05534347
Title: Angiogenic Inflammatory Biomarkers in Juvenile Idiopathic Arthritis
Brief Title: Angiogenic Biomarkers in Juvenile Idiopathic Arthritis
Acronym: MAJIC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220364; 2022-A00468-35 (Other: France : ANSM)
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: Juvenile idiopathic arthritis (JIA); JIA patients in transition towards adult ward; Prognosis of JIA; Severity and structural damage in JIA; Angiogenic and inflammatory biomarkers; Semaphorin (SEMA4A), CCN1; Serum fluid; Synovial fluid
MeSH Terms: conditions — Arthritis, Juvenile; Cone-Rod Dystrophy 10; Cornea Plana 1 | interventions — Blood Specimen Collection; Arthrocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Serum samples
  * Synovial fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Juvenile Idiopathic Arthritis: Patients seen in a specialized rheumatology consultation for the management of juvenile idiopathic arthritis in an adult service, after information and collection of their non-opposition.
  Interventions: Biological: Blood sample; Biological: Joint puncture

INTERVENTIONS:
Biological: Blood sample — Addtional tube of blood needed for follow up of patients
Biological: Joint puncture — Joint puncture if needed according to routine care of the patients

SUMMARY:
The aim of the study is to determine whether serum inflammatory angiogenic markers (eg, semaphorins, CCN1) predict severity of juvenile idiopathic arthritis defined by structural progression and/or therapeutic escalation.

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis (JIA) is a heterogeneous group of chronic inflammatory rheumatic diseases beginning before the age of 16. The most common pediatric rheumatologic disease. JIA is the most common pediatric rheumatologic disease. Apart from clinical features and the biological inflammatory syndrome, no predictive parameter for the severity of JIA, especially polyarticular JIA, has been identified. The team has been interested in the prognosis of RA for many years. Thus, the investigators have conducted various studies in search of biological parameters associated with the joint prognosis of RA patients, which allowed the investigator to discover the interest of angiogenic and inflammatory biomarkers such as semaphorins and CCN1 protein. This has been demonstrated in vitro but also in vivo from sera of RA patients. These markers are associated with activity and structural damage in RA.

The project aims to study the interest of these same angiogenic biomarkers in the serum of JIA patients in order to establish whether, as in RA, they are also associated with disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 16 years-old
* Diagnosis of Juvenile Idiopathic Arthritis with specialized follow up in Rheumatology at Cochin Hospital
* No-opposition to the research
* Patient with health insurance
* Mastery of the French language

Exclusion Criteria:

* Patient under curatorship or guardianship
* Patient receiving french state medical aid

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients over (or egal) 16 years old with diagnosis of Juvenile Idiopathic Arthritis starting their follow up in adult rheumatology ward in Cochin hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Dosage of angiogenic markers | 5 years
  Dosage of angiogenic markers by ELISA method in serum. Determine if angiogenic and inflammatory biomarkers are predictive of a more severe disease as reflected by structural joint damage and treatments received.
  Activity measured with questionnaires, and treatments received. Structural damage determined by x-rays during follow up.
Dosage of angiogenic markers | 5 years
  Dosage of angiogenic markers by ELISA method in synovial fluid if available. Determine if angiogenic and inflammatory biomarkers are predictive of a more severe disease as reflected by structural joint damage and treatments received.
  Activity measured with questionnaires, and treatments received. Structural damage determined by x-rays during follow up.
Dosage of inflammatory markers by ELISA method | 5 years
  Dosage of inflammatory markers by ELISA method in serum. Determine if angiogenic and inflammatory biomarkers are predictive of a more severe disease as reflected by structural joint damage and treatments received.
  Activity measured with questionnaires, and treatments received. Structural damage determined by x-rays during follow up.
Dosage of inflammatory markers by ELISA method | 5 years
  Dosage of inflammatory markers by ELISA method in synovial fluid if available. Determine if angiogenic and inflammatory biomarkers are predictive of a more severe disease as reflected by structural joint damage and treatments received.
  Activity measured with questionnaires, and treatments received. Structural damage determined by x-rays during follow up.

SECONDARY OUTCOMES:
Questionnaires | 5 years
  Severity of JIA
Collection of treatments received | 5 years
  Severity of JIA
Structural damage determined by x-rays | 5 years
  Structural damage determined by x-rays during follow up.
Angiogenic biomarkers | At inclusion
  Determine if sera angiogenic biomarkers are associated with clinical subtypes of JIA.
Inflammatory biomarkers | At inclusion
  Determine if sera inflammatory biomarkers are associated with clinical subtypes of JIA.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick ALLANORE, PD, PhD, Principal Investigator — Cochin Hospital, Assistance Publique des Hôpitaux de Paris (AP-HP)
Locations (1):
- Rheumatology Department, Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No